CLINICAL TRIAL: NCT00164359
Title: A Double-blind Randomised Trial to Assess the Tolerability of Amodiaquine Plus Artesunate (AQ-Art) Versus Chlorproguanil Plus Dapsone Plus Artesunate (CDA) in the Treatment of Uncomplicated P. Falciparum Malaria in Malawi
Brief Title: Amodiaquine Plus Artesunate Versus Lapdap Plus Artesunate in the Treatment of Uncomplicated P. Falciparum Malaria in Malawi
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Ministry of Health and Population, Malawi (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDC-NCID-4538; PA#04018
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: Malaria, Falciparum
Keywords: malaria, falciparum; antimalarials
MeSH Terms: conditions — Malaria, Falciparum | interventions — Amodiaquine; Artesunate; chloroguanil, dapsone drug combination

INTERVENTIONS:
Drug: Amodiaquine plus artesunate
Drug: chlorproguanil-dapsone plus artesunate

SUMMARY:
Sulfadoxine-pyrimethamine is the current first-line therapy for uncomplicated malaria in Malawi. Significant resistance of the P. falciparum malaria parasite to this drug has led to an imminent need for the government of Malawi to identify a new first-line therapy for uncomplicated malaria and to implement that new therapy as policy. This protocol is the second of two protocols whose combined purpose is to provide efficacy and side effect data on four antimalarial drug combinations that are candidates for the next first-line therapy for uncomplicated malaria in Malawi. This protocol aims to assess the acceptability and tolerability of amodiaquine in Malawi. It is a double-blind study comparing amodiaquine plus artesunate (AQ-Art, one of the candidate combination therapies) to chlorproguanil/dapsone plus artesunate (CD-Art, another of the candidate combination therapies) in persons 5 years and older, to see if there is a higher incidence of abdominal pain and/or refusal to take the therapy in the AQ-Art group. Amodiaquine was removed from the Malawian national drug registry in 1995 because of a perceived association with abdominal pain. Although no studies were conducted to substantiate this, consensus among clinicians was that patients were refusing amodiaquine with increasing frequency, citing abdominal pain as the reason, so the drug was removed from the registry. Results from this study, along with the efficacy data from the sister protocol in children under five years of age, will help guide the National Malaria Control Program of Malawi in selecting their next first-line antimalarial therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age five years or older
* Axillary temperature >= 37.5 degrees Celsius
* Monoinfection with P. falciparum
* Parasitemia between 2000 and 200000 parasites/microliter
* Hemoglobin concentration >= 7g/dl
* Consent by the patient of patient's adult guardian
* Residence in the locality and willingness to attend for scheduled visits
* Negative urine pregnancy test in women age twelve years and older

Exclusion Criteria:

* Signs of severe or complicated malaria
* altered consciousness
* convulsions
* prostration (inability to sit/stand/suck/drink)
* respiratory distress or breathlessness
* jaundice
* abnormal breathing
* hemoglobinuria
* circulatory collapse
* persistent vomiting (cannot keep down liquids)
* evidence of a diagnosis other than malaria on physical examination
* presence of mixed infection
* presence of severe malnutrition (as evidenced by symmetrical edema involving at least the feet, light hair color, or cachexia)
* contraindications to the antimalarial drugs used, especially history of allergy
* history of receiving a drug with antimalarial activity in the week prior to enrollment

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 212
Dates: Start 2005-04; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Incidence of abdominal pain on days 1, 2, and 3 in the two treatment groups

SECONDARY OUTCOMES:
Rate of adequate clinical and parasitological response at 14 days
Rate of adequate clinical and parasitological response at 28 days
Mean percent change in blood haemoglobin concentration between day 0 and day 28
Incidence of adverse events other than abdominal pain during the period of observation
Rate of Early Treatment Failure (per WHO definition)
Rate of Late Clinical Failure (per WHO definition)
Rate of Late Parasitological Failure (per WHO definition)
Percent of patients with a decrease in haemoglobin concentration
Percent of patients with a decrease in haemoglobin concentration of >= 2g/dl
Prevalence of parasitemia on Day 2
Prevalence of parasitemia on Day 3
Gametocyte prevalence on Day 14
Gametocyte prevalence on day 28

CONTACTS AND LOCATIONS:
Overall Officials: Rachel N Bronzan, MD, MPH, Principal Investigator — Centers for Disease Control and Prevention
Locations (3):
- Malawi (3):
  - Kawale Health Center, Lilongwe, Lilongwe District
  - Machinga District Hospital, Liwonde, Machinga District
  - Matiki Health Center, Dwangwa, Nkhotakota District